CLINICAL TRIAL: NCT05407857
Title: Taiwan Geriatric Study for Dementia Risk Prevention and Cognitive Enhancement by Multi-modal Intervention (TaiPEI)
Brief Title: Taiwan Geriatric Study for Dementia Risk Prevention and Cognitive Enhancement by Multi-modal Intervention
Acronym: TaiPEI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chun Kuan, Physician, Department of Neurology, Principal Investigator, Associate Professor, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202112075
Record Dates: First submitted 2022-01-31; First posted 2022-06-07 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Three groups (on site intervention group, remote intervention group, and control group)
Who Masked: Outcomes Assessor
Masking Description: We will avoid all the outcomes assessors knowing the allocation and intervention groups.
  The participant will only know what treatment is applied until the start of the intervention. We will also suggest the participants not to discuss their interventions and restrict the chance of communication between different intervention groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- On-site (Experimental): The on-site multi-modal intervention will be actively involved in management with nutrition, exercise and cognitive programs. The on-site intervention group requires subjects to participate in prescribed place according to the protocol.
  Interventions: Behavioral: multi-modal non-pharmacological intervention
- Remote (Active Comparator): The remote intervention group is designed for reducing the chances of person-to-person contact response to the current COVID-19 pandemic and development of digital internet. It uses innovative technology combining wearable devices with inertial measurement units, blue-tooth equipment, apps, feedback technology and artificial intelligence based remote comprehensive training programs.
  Interventions: Behavioral: multi-modal non-pharmacological intervention
- Control (Placebo Comparator): The control group will also receive the same health evaluation and education as all intervention groups.
  Interventions: Behavioral: multi-modal non-pharmacological intervention

INTERVENTIONS:
Behavioral: multi-modal non-pharmacological intervention — multi-modal non-pharmacological intervention including the management with nutrition, exercise and cognitive programs

SUMMARY:
A 3-arm randomized controlled trial of multi-modal non-pharmacological Intervention for preventing the risk of dementia in Taiwanese geriatric people

DETAILED DESCRIPTION:
This project proposes an intervention program for dementia prevention based on the Taiwanese model. The investigator(s) will screen the elderly who are not yet demented but are at high risk of dementia and will randomly allocate them into three groups (on site intervention group, remote intervention group, and control group) for a two-year multi-modal non-pharmacological intervention. All intervention groups will be actively involved in management with nutrition, exercise and cognitive programs. The on-site intervention group requires subjects to participate in prescribed place according to the protocol. The remote intervention group is designed for reducing the chances of person-to-person contact response to the current coronavirus disease 2019 (COVID-19) pandemic and development of digital internet. It uses innovative technology combining wearable devices with inertial measurement units, blue-tooth equipment, apps, feedback technology and artificial intelligence based remote comprehensive training programs. During the study period, each group will be regularly monitored the changes of cardiovascular risk factors, physical performance and cognitive function. The results of multimodal intervention mainly from Taipei and New Taipei City will establish the Taiwan FINGER model (TaiPEI) and will have the information of the conditions and feasibility achieved in Taiwan and implementation suggestions in the face of the epidemic. It can be subsequently applied to the brain/body health care institution and to the prevention of dementia and cardiovascular disease of elderly.

ELIGIBILITY:
Inclusion Criteria:

1. People over 60 without dementia
2. Agree to join the study and sign the consent form
3. The Modified Rankin Scale (MRS) scores between 0-1 points
4. Education level: elementary or higher education (6 years) or can read and write Chinese
5. Very early dementia screening scale (AD-8) < 2, or more than 2 points but without dementia diagnoses after refer to a neurologist.
6. Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) Risk Score: above 8; diagnosed with mild cognitive impairment (MCI) or subjective cognitive decline (SCD) in the past six months.

Exclusion Criteria:

1. Have been diagnosed with any kind of dementia
2. Suspected dementia patients or others who are not suitable to participate in the research assessed by a doctor at the first visit
3. Diseases affecting the safety of various interventional activities (such as remaining life less than two years, symptomatic heart/cerebrovascular disease within 6 months, vascular reperfusion or reconstruction-related surgery within one year, etc., malignant tumor within one year)
4. Severe blindness, hearing or communication impairment, or other difficulty in cooperating or completing assessments and interventions (especially exercise) in the study
5. Severe mental illnesses, including major depression disorder, or major neuromusculoskeletal disorders that are not suitable to join the study.
6. Drug or alcohol abuse in the last year
7. Overlapping with other interventional trials at the same time which may affect the evaluation results.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognition including individual cognitive domains, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  A composite z-score will be obtained from the neuropsychological tests evaluating multiple cognitive domains, including memory, language, process speed, visuospatial, and executive function.

SECONDARY OUTCOMES:
Change in physical assessment, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Senior Fitness Test (SFT) measures six functional areas of physical function (strength, endurance, balance, agility, and flexibility)
Change in physical assessment, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Short Physical Performance Battery (SPPB), score range: 0-12; higher scores mean a better outcome.
Change in physical assessment, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  International Physical Activity Questionnaire (IPAQ), a 27-item self-reported measure of physical activity
Change in physical functioning - Hand-grip strength, kg | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Measured using a hand-grip dynamometer
Change of the questionnaire regarding the nutrition, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Mini Nutritional Assessment-Short Form (MNA-SF), a screening scale used to assess current nutritional status. score range: 0-14, higher scores mean a better outcome.
Change of the questionnaire regarding the nutrition, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  food frequency questionnaire (FFQ), a finite list of foods and beverages with response categories to indicate usual frequency of consumption over the time period
Change of nutrition intake, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  3-day dietary record: a self-reported account of all foods and beverages consumed within recent three days
Change in functioning level, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Activities of Daily Living Questionnaire (ADLQ)
Change in functioning level, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  The Brief University of California San Diego (UCSD) Performance-Based Skills Assessment (UPSA-Brief) -Traditional Chinese Version: two subdomains (Finances, Communication) with a total score ranging from 0 to 100.
Change in functioning level, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Florida Cognitive Activities Scale (FCAS): a 25-item scale used to assess cognitive activities in the elderly with two subscales (Higher Cognitive Abilities and Frequent Cognitive Abilities)
Change in functioning level, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  EuroQol five-dimensional (EQ-5D): an instrument for measuring quality of life regarding the five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in functioning level, unit on a scale | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Activities of Daily Living Questionnaire (ADLQ), The Brief University of California San Diego (UCSD) Performance-Based Skills Assessment（Traditional Chinese Version）（UPSA-Brief）, Florida Cognitive Activities Scale(FCAS), EuroQol five-dimensional (EQ-5D)
Change in depressive symptoms, unit on a scale. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Geriatric Depression Scale-Short Form (GDS-S), score range: 0-15; higher scores mean a worse outcome.
Change in sleep symptoms, unit on a scale. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Epworth sleepiness scale (ESS)
Change in sleep symptoms, unit on a scale. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Pittsburgh Sleep Quality Index (PSQI)
Change in blood tests - fasting plasma glucose, mmol/L. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Measured from fasting blood sample
Change in blood tests - triglycerides, mmol/L. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Measured from fasting blood sample
Change in blood tests - Albumin, prealbumin, g/dL. | Before intervention (Baseline); During intervention (every six month); follow-up (6 months after intervention ends)
  Measured from fasting blood sample
Change of Plasma amyloid beta, pg/mL | Before intervention (Baseline); During intervention (6th month and 24th month)
  Assessed by ultra-sensitive, immunomagnetic reduction assay (MagQu, LLC, Surprise, AZ),
Change of Plasma tau, pg/mL | Before intervention (Baseline); During intervention (6th month and 24th month)
  Assessed by ultra-sensitive, immunomagnetic reduction assay (MagQu, LLC, Surprise, AZ),

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chun Kuan, MD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, New Taipei City, Taiwan